CLINICAL TRIAL: NCT02852980
Title: Retrospective Study to Estimate Screening of the Type 2 Diabetes of Women Who Had Childbirth in the Hospital Center Rene Dubos and Having Gestational Diabetes
Brief Title: Estimate Rate of the Women Who Have Gestational Diabetes
Acronym: ERD2-DIGERD
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1114
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gestational diabetes women: Women who had childbirth in the Hospital center Rene Dubos and who had gestational diabetes.
  Interventions: Other: gestational diabetes women

INTERVENTIONS:
Other: gestational diabetes women — No intervention.

SUMMARY:
Retrospective study to estimate screening of the type 2 diabetes of women who had childbirth in the Hospital center Rene Dubos and having gestational diabetes.

DETAILED DESCRIPTION:
It is recognized that pregnant women who had gestational diabetes (DG) multiplied by 7 subsequent risk of developing type 2 diabetes and this during 25 years. There is at present no formal recommendation of the High Authority for Health (HAS) as an organization of a long term screening for those women. However the recommendations of CNGOF (French Council of Gynaecologists and Obstetricians) and SFD (French society of diabetes) recommend screening for type 2 diabetes after a gestational diabetes in the postnatal consultation. But today how many women views due to a gestational diabetes have realized their screening? It is likely that the rate of occurrence of type 2 diabetes after gestational diabetes is underestimated today. Otherwise it is possible that the occurrence of type 2 diabetes is associated with some risk factors such as high BMI, insulin therapy during pregnancy. Another interrogation is the role of the doctor to reduce the number of women who do not realize their screening at 3 months postpartum. Better awareness of the importance of long term monitoring would reduce the proportion of women who do not realize their screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged over 18 years
* Participants who deliver between 01/01/2013 and 30/06/2015
* Participants who have had a gestational diabetes
* Participants who have been informed and have returned the questionary

Exclusion Criteria:

* Participants who do not wishing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who had childbirth in the Hospital center Rene Dubos and having gestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Glycemia realized after childbirth | 3 months
  The investigators want to know the number of women who realized a Glycemia analysis.

SECONDARY OUTCOMES:
Percentage of women who have pursued the dietary and hygiene rules | 3 months
  Information about dietary and hygiene rules are collected on a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CAMPINOS, PH, Principal Investigator — Rene Dubos Hospital
Locations (1):
- Rene Dubos Hospital, Pontoise, Val d'Oise, France

IPD SHARING:
Plan to Share IPD: No